CLINICAL TRIAL: NCT03539588
Title: Trigger Point Dry Needling vs Trigger Point Dry Needling With Intramuscular Electrical Stimulation for the Treatment of Sub-acute and Chronic Low Back Pain in a Military Population: A Randomized Crossover Design
Brief Title: Trigger Point Dry Needling vs Trigger Point Dry Needling With Intramuscular Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-26
Record Dates: First submitted 2017-03-10; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Sub-acute and Chronic Low Back Pain
Keywords: dry needling; electrical stimulation; E-Stim; LBP; low back pain; trigger point; chronic; subacute
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group 1 (Active Comparator): In this group participants will receive trigger point dry needling with electrical stimulation first and receive trigger point needling by itself second. Only MYOTECH dry needles will be used in this study. However we are not studying the equipment.
  Interventions: Device: trigger point dry needling; Device: Electrical Stimulation
- Treatment Group 2 (Active Comparator): In this group the participants will receive trigger point dry needling first and receive trigger point dry needling with electrical stimulation second. Only MYOTECH dry needles and ESTIM II dual channel stimulator will be used in this study. However we are not studying the equipment.
  Interventions: Device: trigger point dry needling; Device: Electrical Stimulation

INTERVENTIONS:
Device: trigger point dry needling — placement of the dry needle into the muscle tissue to elicit a local twitch response. Only MYOTECH dry needles and ESTIM II dual channel stimulator will be used in this study. However we are not studying the equipment.
Device: Electrical Stimulation — uses the dry needles as nodes to stimulate muscular contraction. Only MYOTECH dry needles and ESTIM II dual channel stimulator will be used in this study. However we are not studying the equipment.

SUMMARY:
trigger point dry needling with intramuscular electrical stimulation vs trigger point dry needling

DETAILED DESCRIPTION:
The purpose of this study is to evaluate if trigger point dry needling with intramuscular electrical stimulation is more effective in decreasing pain and disability in individuals with sub-acute and chronic low back pain (LBP) than with trigger point dry needling alone. The investigators are using a within subjects randomized crossover study that will recruit 30 active duty military personnel or beneficiaries from William Beaumont Army Medical Center and all associated clinics. The investigators hypothesize that individuals with LBP will exhibit larger improvements in pain and disability when receiving trigger point dry needling with intramuscular electrical stimulation than when receiving trigger point dry needling alone.

ELIGIBILITY:
Inclusion Criteria:

* Currently experience low back pain for greater than 4 weeks (Low back pain defined as pain below the T12th vertebrae with or without radiation) Military or DOD Beneficiary (any branch; 18-65 years of age)

Exclusion Criteria:

* Structural Deformity (ankylosing Spondylitis, Scoliosis)
* Has any other Orthopedic condition that may keep subject from performing Low - Back Exercises
* Tumors
* Spinal infection or local infection
* Pregnancy-All female subjects will be given either a blood serum or urine pregnancy test.
* Spinal cord compression or Cauda Equina Syndrome
* Subject with the inability to keep appointments
* Has History of prior surgery
* Has received Dry Needling or Acupuncture in the last 6 months
* History of bleeding disorders
* High anti-coagulant use
* History of immune suppression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale to assess change | Baseline and before and after each treatment session, duration per subject is approximately 3 weeks
  an 11 point scale on which the participant will grade their pain

CONTACTS AND LOCATIONS:
Overall Officials: David K Hulsizer, DPT, Principal Investigator — WBAMC
Locations (1):
- William BAMC, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armed Forces Health Surveillance Center-AFHSC. Absolute and relative morbidity burdens attributable to various illnesses and injuries, U.S. Armed Forces, 2011. MSMR. 2012 Apr;19(4):4-8; discussion 8-9. No abstract available. PMID 22587833
- [Background] April 2012 - v19_n04 - v19_n04.pdf." Accessed May 18, 2016. https://www.afhsc.mil/documents/pubs/msmrs/2012/v19_n04.pdf#Page=2.
- [Background] Brinkhaus B, Witt CM, Jena S, Linde K, Streng A, Wagenpfeil S, Irnich D, Walther HU, Melchart D, Willich SN. Acupuncture in patients with chronic low back pain: a randomized controlled trial. Arch Intern Med. 2006 Feb 27;166(4):450-7. doi: 10.1001/archinte.166.4.450. PMID 16505266
- [Background] Cagnie B, Dewitte V, Barbe T, Timmermans F, Delrue N, Meeus M. Physiologic effects of dry needling. Curr Pain Headache Rep. 2013 Aug;17(8):348. doi: 10.1007/s11916-013-0348-5. PMID 23801002
- [Background] Cherkin DC, Sherman KJ, Avins AL, Erro JH, Ichikawa L, Barlow WE, Delaney K, Hawkes R, Hamilton L, Pressman A, Khalsa PS, Deyo RA. A randomized trial comparing acupuncture, simulated acupuncture, and usual care for chronic low back pain. Arch Intern Med. 2009 May 11;169(9):858-66. doi: 10.1001/archinternmed.2009.65. PMID 19433697
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Cohen SP, Brown C, Kurihara C, Plunkett A, Nguyen C, Strassels SA. Diagnoses and factors associated with medical evacuation and return to duty among nonmilitary personnel participating in military operations in Iraq and Afghanistan. CMAJ. 2011 Mar 22;183(5):E289-95. doi: 10.1503/cmaj.100244. Epub 2011 Feb 14. PMID 21324873
- [Background] Cohen SP, Griffith S, Larkin TM, Villena F, Larkin R. Presentation, diagnoses, mechanisms of injury, and treatment of soldiers injured in Operation Iraqi Freedom: an epidemiological study conducted at two military pain management centers. Anesth Analg. 2005 Oct;101(4):1098-1103. doi: 10.1213/01.ane.0000169332.45209.cf. PMID 16192528
- [Background] Cummings TM, White AR. Needling therapies in the management of myofascial trigger point pain: a systematic review. Arch Phys Med Rehabil. 2001 Jul;82(7):986-92. doi: 10.1053/apmr.2001.24023. PMID 11441390
- [Background] Deyo RA, Mirza SK, Martin BI. Back pain prevalence and visit rates: estimates from U.S. national surveys, 2002. Spine (Phila Pa 1976). 2006 Nov 1;31(23):2724-7. doi: 10.1097/01.brs.0000244618.06877.cd. PMID 17077742
- [Background] Deyo RA, Mirza SK, Turner JA, Martin BI. Overtreating chronic back pain: time to back off? J Am Board Fam Med. 2009 Jan-Feb;22(1):62-8. doi: 10.3122/jabfm.2009.01.080102. PMID 19124635
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Eisenberg DM, Post DE, Davis RB, Connelly MT, Legedza AT, Hrbek AL, Prosser LA, Buring JE, Inui TS, Cherkin DC. Addition of choice of complementary therapies to usual care for acute low back pain: a randomized controlled trial. Spine (Phila Pa 1976). 2007 Jan 15;32(2):151-8. doi: 10.1097/01.brs.0000252697.07214.65. PMID 17224808
- [Background] Ernat J, Knox J, Orchowski J, Owens B. Incidence and risk factors for acute low back pain in active duty infantry. Mil Med. 2012 Nov;177(11):1348-51. doi: 10.7205/milmed-d-12-00183. PMID 23198512
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Fritz JM, George SZ. Identifying psychosocial variables in patients with acute work-related low back pain: the importance of fear-avoidance beliefs. Phys Ther. 2002 Oct;82(10):973-83. PMID 12350212
- [Background] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Background] Furlan AD, van Tulder M, Cherkin D, Tsukayama H, Lao L, Koes B, Berman B. Acupuncture and dry-needling for low back pain: an updated systematic review within the framework of the cochrane collaboration. Spine (Phila Pa 1976). 2005 Apr 15;30(8):944-63. doi: 10.1097/01.brs.0000158941.21571.01. PMID 15834340
- [Background] George SZ, Childs JD, Teyhen DS, Wu SS, Wright AC, Dugan JL, Robinson ME. Rationale, design, and protocol for the prevention of low back pain in the military (POLM) trial (NCT00373009). BMC Musculoskelet Disord. 2007 Sep 14;8:92. doi: 10.1186/1471-2474-8-92. PMID 17868436
- [Background] Gilbert FJ, Grant AM, Gillan MG, Vale LD, Campbell MK, Scott NW, Knight DJ, Wardlaw D; Scottish Back Trial Group. Low back pain: influence of early MR imaging or CT on treatment and outcome--multicenter randomized trial. Radiology. 2004 May;231(2):343-51. doi: 10.1148/radiol.2312030886. Epub 2004 Mar 18. PMID 15031430
- [Background] Giles LG, Muller R. Chronic spinal pain: a randomized clinical trial comparing medication, acupuncture, and spinal manipulation. Spine (Phila Pa 1976). 2003 Jul 15;28(14):1490-502; discussion 1502-3. doi: 10.1097/00007632-200307150-00003. PMID 12865832
- [Background] Gunn CC, Milbrandt WE, Little AS, Mason KE. Dry needling of muscle motor points for chronic low-back pain: a randomized clinical trial with long-term follow-up. Spine (Phila Pa 1976). 1980 May-Jun;5(3):279-91. doi: 10.1097/00007632-198005000-00011. No abstract available. PMID 6446774
- [Background] Haake M, Muller HH, Schade-Brittinger C, Basler HD, Schafer H, Maier C, Endres HG, Trampisch HJ, Molsberger A. German Acupuncture Trials (GERAC) for chronic low back pain: randomized, multicenter, blinded, parallel-group trial with 3 groups. Arch Intern Med. 2007 Sep 24;167(17):1892-8. doi: 10.1001/archinte.167.17.1892. PMID 17893311
- [Background] Hart LG, Deyo RA, Cherkin DC. Physician office visits for low back pain. Frequency, clinical evaluation, and treatment patterns from a U.S. national survey. Spine (Phila Pa 1976). 1995 Jan 1;20(1):11-9. doi: 10.1097/00007632-199501000-00003. PMID 7709270
- [Background] Hebert JJ, Koppenhaver SL, Walker BF. Subgrouping patients with low back pain: a treatment-based approach to classification. Sports Health. 2011 Nov;3(6):534-42. doi: 10.1177/1941738111415044. PMID 23016055
- [Background] Heliovaara M, Sievers K, Impivaara O, Maatela J, Knekt P, Makela M, Aromaa A. Descriptive epidemiology and public health aspects of low back pain. Ann Med. 1989 Oct;21(5):327-33. doi: 10.3109/07853898909149216. PMID 2532521
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Hong CZ, Simons DG. Pathophysiologic and electrophysiologic mechanisms of myofascial trigger points. Arch Phys Med Rehabil. 1998 Jul;79(7):863-72. doi: 10.1016/s0003-9993(98)90371-9. PMID 9685106
- [Background] Hsieh YL, Kao MJ, Kuan TS, Chen SM, Chen JT, Hong CZ. Dry needling to a key myofascial trigger point may reduce the irritability of satellite MTrPs. Am J Phys Med Rehabil. 2007 May;86(5):397-403. doi: 10.1097/PHM.0b013e31804a554d. PMID 17449984
- [Background] Inoue M, Kitakoji H, Ishizaki N, Tawa M, Yano T, Katsumi Y, Kawakita K. Relief of low back pain immediately after acupuncture treatment--a randomised, placebo controlled trial. Acupunct Med. 2006 Sep;24(3):103-8. doi: 10.1136/aim.24.3.103. PMID 17013356
- [Background] Jarvik JG, Deyo RA. Diagnostic evaluation of low back pain with emphasis on imaging. Ann Intern Med. 2002 Oct 1;137(7):586-97. doi: 10.7326/0003-4819-137-7-200210010-00010. PMID 12353946
- [Background] Johnston BC, da Costa BR, Devereaux PJ, Akl EA, Busse JW; Expertise-Based RCT Working Group. The use of expertise-based randomized controlled trials to assess spinal manipulation and acupuncture for low back pain: a systematic review. Spine (Phila Pa 1976). 2008 Apr 15;33(8):914-8. doi: 10.1097/BRS.0b013e31816b4be4. PMID 18404113
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] Konitzer LN, Fargo MV, Brininger TL, Lim Reed M. Association between back, neck, and upper extremity musculoskeletal pain and the individual body armor. J Hand Ther. 2008 Apr-Jun;21(2):143-8; quiz 149. doi: 10.1197/j.jht.2007.10.017. PMID 18436136
- [Background] Larsson R, Oberg AP, Larsson SE. Changes of trapezius muscle blood flow and electromyography in chronic neck pain due to trapezius myalgia. Pain. 1999 Jan;79(1):45-50. doi: 10.1016/S0304-3959(98)00144-4. PMID 9928775
- [Background] Lee SH, Chen CC, Lee CS, Lin TC, Chan RC. Effects of needle electrical intramuscular stimulation on shoulder and cervical myofascial pain syndrome and microcirculation. J Chin Med Assoc. 2008 Apr;71(4):200-6. doi: 10.1016/S1726-4901(08)70104-7. PMID 18436503
- [Background] Lewit K. The needle effect in the relief of myofascial pain. Pain. 1979 Feb;6(1):83-90. doi: 10.1016/0304-3959(79)90142-8. PMID 424236
- [Background] Lincoln AE, Smith GS, Amoroso PJ, Bell NS. The natural history and risk factors of musculoskeletal conditions resulting in disability among US Army personnel. Work. 2002;18(2):99-113. PMID 12441574
- [Background] Lucas N, Macaskill P, Irwig L, Moran R, Bogduk N. Reliability of physical examination for diagnosis of myofascial trigger points: a systematic review of the literature. Clin J Pain. 2009 Jan;25(1):80-9. doi: 10.1097/AJP.0b013e31817e13b6. PMID 19158550
- [Background] Lurie JD, Birkmeyer NJ, Weinstein JN. Rates of advanced spinal imaging and spine surgery. Spine (Phila Pa 1976). 2003 Mar 15;28(6):616-20. doi: 10.1097/01.BRS.0000049927.37696.DC. PMID 12642771
- [Background] Manheimer E, White A, Berman B, Forys K, Ernst E. Meta-analysis: acupuncture for low back pain. Ann Intern Med. 2005 Apr 19;142(8):651-63. doi: 10.7326/0003-4819-142-8-200504190-00014. PMID 15838072
- [Background] Molsberger AF, Mau J, Pawelec DB, Winkler J. Does acupuncture improve the orthopedic management of chronic low back pain--a randomized, blinded, controlled trial with 3 months follow up. Pain. 2002 Oct;99(3):579-587. doi: 10.1016/S0304-3959(02)00269-5. PMID 12406534
- [Background] Napadow V, Makris N, Liu J, Kettner NW, Kwong KK, Hui KK. Effects of electroacupuncture versus manual acupuncture on the human brain as measured by fMRI. Hum Brain Mapp. 2005 Mar;24(3):193-205. doi: 10.1002/hbm.20081. PMID 15499576
- [Background] Rainey CE. The use of trigger point dry needling and intramuscular electrical stimulation for a subject with chronic low back pain: a case report. Int J Sports Phys Ther. 2013 Apr;8(2):145-61. PMID 23593553
- [Background] Tough, Elizabeth A., and Adrian R. White. "Effectiveness of Acupuncture/dry Needling for Myofascial Trigger Point Pain." Physical Therapy Reviews 16, no. 2 (2011): 147-54.
- [Background] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479
- [Background] Vas J, Aranda JM, Modesto M, Benitez-Parejo N, Herrera A, Martinez-Barquin DM, Aguilar I, Sanchez-Araujo M, Rivas-Ruiz F. Acupuncture in patients with acute low back pain: a multicentre randomised controlled clinical trial. Pain. 2012 Sep;153(9):1883-1889. doi: 10.1016/j.pain.2012.05.033. Epub 2012 Jul 4. PMID 22770838
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Witt CM, Pach D, Brinkhaus B, Wruck K, Tag B, Mank S, Willich SN. Safety of acupuncture: results of a prospective observational study with 229,230 patients and introduction of a medical information and consent form. Forsch Komplementmed. 2009 Apr;16(2):91-7. doi: 10.1159/000209315. Epub 2009 Apr 9. PMID 19420954
- [Background] Yeung CK, Leung MC, Chow DH. The use of electro-acupuncture in conjunction with exercise for the treatment of chronic low-back pain. J Altern Complement Med. 2003 Aug;9(4):479-90. doi: 10.1089/107555303322284767. PMID 14499023